CLINICAL TRIAL: NCT03694496
Title: A Randomized Controlled Trial Evaluating the Efficacy of a Peer-led Theory-based Intervention in Promoting Healthy Behaviors Among Adolescents in Hong Kong
Brief Title: The Effectiveness of an Oral Health Education Programme of Adolescents in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UW 18-029
Record Dates: First submitted 2018-09-19; First posted 2018-10-03 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-02

CONDITIONS: Caries, Dental; Periodontal Diseases
MeSH Terms: conditions — Dental Caries; Periodontal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: .An experienced fieldworker will facilitate the survey process, and she will be blind to our group allocation. Two experienced dentists will conduct the dental examinations who don't know the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peer-led theory-based intervention group (Experimental): 2-6 students (depending on the headcount of the grade 2 students of the school) will be selected as peer leaders and they will receive oral health training first. After being trained and qualified, they will deliver oral health talks and workshops to their peers. The peer leaders will be requested to conduct six activities during 6 months, including health talks, workshops, information leaflets, etc.
  Interventions: Behavioral: peer-led theory-based intervention group
- Control group (No Intervention): Participants in the control group will continue their present practice, and no additional interventions will be given except oral health pamphlets delivery. We will record their present practice in detail. As the control group is in different schools, so they will have very low opportunity to get access to the peer-led activities conducted in the intervention group. Contamination will be quite minimum.

INTERVENTIONS:
Behavioral: peer-led theory-based intervention group — We plan to select 2-8 peer leaders in S2 students within each school in the intervention group. A total of 25-48 peer leaders will be selected and trained in this study.
  An experienced behavioural scientist will train the peer leaders through lectures, workshops, and individual counselling.
  A total of 6 hours training (3 hours per day x 2 days) will be conducted during weekends. Peer leaders will practice in groups, and only those who pass the evaluation are allowed to conduct peer-led interventions. We will record the performance and give specific feedback to each peer leader.
  Arms: peer-led theory-based intervention group

SUMMARY:
This project aims to evaluate the relative efficacy of a peer-led intervention based on the Social Cognitive Theory and Health Belief Model versus the control (only pamphlet delivery) on increasing the prevalence of healthy oral behaviors and oral health status among adolescents in Hong Kong. A two-arm non-blinded randomized controlled trial will be conducted among random samples of adolescents enrolling in secondary schools in Hong Kong. In addition to a baseline survey, two follow-up evaluative surveys will be conducted at months 6 and 12. Survey questionnaires will be conducted to participants at three time points (baseline, 6-, 12-month follow-up). Dental check-up examinations will be evaluated at two time points (baseline, 6-month follow-up). Repeated measures will be used to record participants' background, oral behaviors, theory based cognition, and potential confounders. Validated scales will be used. DMFT, plaque index and CPI index will be used to assess the oral health status of participants.

DETAILED DESCRIPTION:
Baseline survey and dental examination The baseline survey will collect information on participants' background characteristics (e.g., socio-demographics), Social Cognitive Theory (SCT)-related variables (perceived susceptibility, perceived severity, perceived benefits, perceived barriers, self-efficacy), Health Belief Model (HBM)-related variables (reciprocal determinism, behavioral capability, outcome expectations), and oral health behaviors. Validated scales have been identified and will be used in the survey.

To comprehensively assess each participant's oral health status at baseline, their oral hygiene status, caries experience and periodontal condition will be recorded following the recommendations of the World Health Organization (WHO) for oral health surveys. Oral hygiene status will be recorded through plaque index (PI) (Quigley Hein, 1972) on a scale of 0 to 5. Dental caries experience will be recorded by counting the numbers of permanent teeth that are decayed (DT), missing due to caries (MT), and filled (FT) to generate a DMFT score. Periodontal condition will be recorded using the Community Periodontal Index (CPI). Two trained and calibrated examiners (kappa = 0.81 - 0.87 for intra- and inter-examiner reliabilities for the assessment of DMFT and CPI) will perform the clinical examinations using a plane disposable plane intra-oral mirror with a built-in LED light source and a WHO CPI periodontal probe. Ten percent of the participants will be randomly selected and re-examined in each school to continuously monitor intra- and inter-examiner reliabilities of assessing PI DMFT and CPI.

Intervention description A total of five peer-led activities will be conducted in the intervention schools by the well-trained peer leaders within a 6-month intervention period.

1. In the 1st month of intervention, peer leaders will deliver a poster and a leaflet providing information on healthy oral behaviors based on SCT and HBM. Such materials will be provided at the entrance of the school gate, the canteen, and each class. Peer leaders will encourage students to ask questions when they receive such materials. Participants are free to take an on-site quiz to check assess their knowledge level.
2. In the 2nd month of intervention, peer leaders will give a specific health talk aiming to raise the awareness of healthy oral behaviors. Schools teachers will encourage all students to participate in this talk. We will video-record this health talk and make it available online to reach more students. This talk will be guided by SCT and HBM, and it will include short testimonials of the good experiences of the peer leaders when performing healthy oral behaviors.
3. In the 3rd month of intervention, peer leaders will organize a workshop aiming to help the participants practicing skills in performing healthy oral behaviors. Regarding different oral behaviors (tooth brushing, dental flossing, and dental visits), targeted skills will be practiced.
4. In the 4th month of intervention, peer leaders are encouraged to self-design and conduct one more oral health-related activity that they are interested. Necessary support will be provided by the team. We will record details of this peer leader-initiated activity.
5. In the 5th or 6th month of intervention, peer leaders will deliver a special talk regarding illness representations for students with existing oral diseases only. The talk will focus on improving illness representation in both cognitive and emotional aspects, and coping strategies will be practiced.

The first follow-up at months 6 The first follow-up at months 6 will include two parts. The first part is to collect participants' self-reported data through questionnaire. An experienced fieldworker will facilitate the survey process, and she will be blind to our group allocation. The month 6 follow-up data suggest an immediate impact of the intervention, as all intervention activities will be conducted within this 6-month intervention period. The proposed time interval (6 months) is reasonable and feasible, as 6 months is the most frequently adopted time frame to assess behavior changes and the dental visit for check-up (one of our primary outcomes) is recommended to adolescents every 6 months. We will compare changes before and after this intervention within interventions group, and we will also investigate the differences between intervention group and control group.

The second follow-up at months 12 The second follow-up at months 12 will include two parts. The first part is to collect participants' self-reported data through survey, the same procedure as the first follow-up at month 6. The month 12 follow up data suggest a prolonged impact of the intervention, as no intervention activities will be conducted between months 6 and months 12.

The second part is to do dental re-examination, using the same methods and criteria as the baseline examination. We will compare the disease status changes before and after intervention within interventions group. The consistency between self-reported healthy oral behaviors and dental examination outcomes will also be calculated. No dental examination will be conducted at month 6 follow up, as oral disease status is not likely to change within a short time period like 6 months.

Data analysis The intra- and inter-examiner reliabilities of assessing PI, DMFT and CPI at the tooth level will be tested through the use of the kappa statistic. Data of DMFT and CPI at the tooth level will be used to generate the oral disease status at the subject level.

Intention-to-treat analysis will be conducted. Multiple imputation methods will be used to deal with missing data if it occurs. Between-group (intervention versus control) baseline differences in the frequency distributions of potential confounders will be compared by using chi-square test, t-test, Mann-Whitney test or other statistics. The absolute and relative risks and number needed to treat (and their 95% confidence intervals) for the binary outcomes comparing the two groups at months 6 and 12 will be derived. Adjusted comparisons between the intervention and control groups will be made for all binary outcomes, adjusting for any potential confounders showing p<.10 in the between-group baseline comparisons (if any), using modified Poisson regression with robust sandwich variance estimation. SPSS will be used for data analysis; p<.05 (2-sided) will be taken as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2 students of Secondary schools at the baseline recruitment
* Agree to voluntarily participate
* Do not intend to leave Hong Kong within the next 12 months

Exclusion Criteria:

* undergoing orthondontic treatment

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1184 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Oral health behaviors | 12 months
  It was evaluated using a self-report measure. Tooth brushing, flossing will be aluated by asking how often you performed this behavior. The answer should be two times a day, once a day, several times per week, once a week, never.

SECONDARY OUTCOMES:
Cognition related to oral health knowledge | 12 months
  The three components of the HBM constructs and two components of SCT were measured using a self-reported questionnaire. Cronbach's alpha coefficients were 0.74, 0.84, 0.86 for items of HBM and 0.96, 0.74 for items of SCT. Item-total and item-subscale correlation coefficients were also satisfactory (ranging from 0.62 to 0.94, all p<0.05). All the constructs were measured by 59 items. Item responses were measured on a five-point Likert scale; responses ranged from 1 (strongly disagree) to 5 (strongly agree). The average score will be calculated (ranging from 1 to 5). Higher score represents a lower cognition of psychological constructs.
Child Oral Health Quality of Life Questionnaire (CPQ-16) | 12 months
  Child oral health quality of life was evaluated by 16 items. The response options for each item were "never" (scoring 1), "once or twice" (scoring 2), "sometimes" (scoring 3), "often" (scoring 4), or "every day or almost every day (scoring 5). Cronbach's alpha coefficient of this scale was 0.89. The mean inter-item correlations ranged from 0.68 (oral symptoms) to 0.88 (social well-being). The total score of all the items will be calculated (ranging from 16-80). Higher scores represents a lower oral health related quality of life
Oral health knowledge assessment | 12 months
  To assess adolescents' dental knowledge, 21 multiple choice questions on the cause and prevention of dental diseases were asked. One point was given to each correct answer; and no point was given to a wrong answer or a 'don't know' answer. Thus, the dental knowledge score could range from 0 to 21. The adolescents were then categorized into three groups according to their dental knowledge scores - poor (scored 0-7), moderate (scored 8-14) and good (scored 15-21).
Modified Child Dental Anxiety Scale (MCDAS) | 12 months
  Dental anxiety of adolescents was evaluated by 8 items. Each question was answered by using five-Likert scale (not worried=1; very slightly worried=2; fairly worried=3; worried a lot=4; very worried=5). The range of the score was 8-40. Higher scores indicate a more severe dental anxiety.
Generalized Anxiety Disorder-7 (GAD-7) | 12 months
  GAD-7 was used to evaluate generalized anxiety of adolescents. It was a seven-item self-rating instrument. Each item described one of the typical symptoms of GAD and was evaluated by the frequency in which that symptom emerged over the last two weeks: "Not at all" scored 0, "Several days" scored 1, "More than half the days" scored 2, and "Nearly every day" scored 3. The total score range from 0-21. Higher score indicates a more severe generalized anxiety.
Self-percept Social Support | 12 months
  Material support and emotional support provided from family members, friends and teachers were asked .It was grade using 0-10 point, "0" means "no support", "10" means "a lot of support". The value of each item would be evaluated separately. Lower score means poorer support, higher score means better support.
Plaque Index (Quigley Hein, 1972) | 12 months
  An index that evaluates the plaque revealed on the buccal non-restored surfaces of the teeth on a scale of 0 to 5, defined by G. A. Quigley and J. W. Hein in 1962 and modified by S. Turesky, N. D. Gilmore, and I. Glickman in 1970. All teeth except the third molars are assessed. An index for the entire mouth is determined by dividing the total score by the number of surfaces examined.
  Quigley-Hain plaque index 0-No plaque
  1. Isolated flecks of plaque at the gingival margin
  2. A continuous band of plaque up to 1mm at the gingival margin
  3. Plaque greater than 1mm in width and covering up to one third of the tooth surface
  4. Plaque covering from one thirds to two thirds of the tooth surface
  5. Plaque covering more than two thirds of the tooth surface
DMFT (WHO, 5th edition) | 12 months
  DMFT (number of Decayed, Missing due to caries, and Filled Teeth in the permanent dentition)

CONTACTS AND LOCATIONS:
Overall Officials: Hai Ming WONG, PhD, Principal Investigator — the Faculty of Dentistry, The University of Hong Kong
Locations (1):
- the Faculty of Dentistry, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen PE. [Continuous improvement of oral health in the 21st century: the approach of the WHO Global Oral Health Programme]. Zhonghua Kou Qiang Yi Xue Za Zhi. 2004 Nov;39(6):441-4. No abstract available. Chinese. PMID 15854309
- [Background] Shaw WC, Meek SC, Jones DS. Nicknames, teasing, harassment and the salience of dental features among school children. Br J Orthod. 1980 Apr;7(2):75-80. doi: 10.1179/bjo.7.2.75. No abstract available. PMID 6932969
- [Background] McGrath C, Broder H, Wilson-Genderson M. Assessing the impact of oral health on the life quality of children: implications for research and practice. Community Dent Oral Epidemiol. 2004 Apr;32(2):81-5. doi: 10.1111/j.1600-0528.2004.00149.x. PMID 15061856
- [Background] Mak KK, Day JR. Dental health behaviours among early adolescents in Hong Kong. Int J Dent Hyg. 2011 May;9(2):122-6. doi: 10.1111/j.1601-5037.2010.00452.x. PMID 21078081
- [Background] Wong HM, McGrath CP, King NM, Lo EC. Oral health-related quality of life in Hong Kong preschool children. Caries Res. 2011;45(4):370-6. doi: 10.1159/000330231. Epub 2011 Aug 3. PMID 21822015
- [Background] de Silva AM, Hegde S, Akudo Nwagbara B, Calache H, Gussy MG, Nasser M, Morrice HR, Riggs E, Leong PM, Meyenn LK, Yousefi-Nooraie R. Community-based population-level interventions for promoting child oral health. Cochrane Database Syst Rev. 2016 Sep 15;9(9):CD009837. doi: 10.1002/14651858.CD009837.pub2. PMID 27629283
- [Background] Watt RG. Strategies and approaches in oral disease prevention and health promotion. Bull World Health Organ. 2005 Sep;83(9):711-8. Epub 2005 Sep 30. PMID 16211164
- [Background] Wu L, Gao X, Lo ECM, Ho SMY, McGrath C, Wong MCM. Motivational Interviewing to Promote Oral Health in Adolescents. J Adolesc Health. 2017 Sep;61(3):378-384. doi: 10.1016/j.jadohealth.2017.03.010. Epub 2017 May 19. PMID 28532895
- [Background] Husseini A, Slot DE, Van der Weijden GA. The efficacy of oral irrigation in addition to a toothbrush on plaque and the clinical parameters of periodontal inflammation: a systematic review. Int J Dent Hyg. 2008 Nov;6(4):304-14. doi: 10.1111/j.1601-5037.2008.00343.x. PMID 19138181
- [Background] Dumitrescu AL, Dogaru BC, Duta C, Manolescu BN. Testing five social-cognitive models to explain predictors of personal oral health behaviours and intention to improve them. Oral Health Prev Dent. 2014;12(4):345-55. doi: 10.3290/j.ohpd.a31662. PMID 24624388
- [Background] Pakpour AH, Sniehotta FF. Perceived behavioural control and coping planning predict dental brushing behaviour among Iranian adolescents. J Clin Periodontol. 2012 Feb;39(2):132-7. doi: 10.1111/j.1600-051X.2011.01826.x. Epub 2011 Dec 12. PMID 22150555
- [Background] Mellanby AR, Rees JB, Tripp JH. Peer-led and adult-led school health education: a critical review of available comparative research. Health Educ Res. 2000 Oct;15(5):533-45. doi: 10.1093/her/15.5.533. PMID 11184213
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Janz NK, Becker MH. The Health Belief Model: a decade later. Health Educ Q. 1984 Spring;11(1):1-47. doi: 10.1177/109019818401100101. PMID 6392204
- [Derived] Xiang B, Wong HM, McGrath CPJ. The efficacy of peer-led oral health programs based on Social Cognitive Theory and Health Belief Model among Hong Kong adolescents: a cluster-randomized controlled trial. Transl Behav Med. 2022 Mar 17;12(3):423-432. doi: 10.1093/tbm/ibab142. PMID 34791503
- [Derived] Xiang B, McGrath CPJ, Wong HM. The Efficacy of a Multi-Theory-Based Peer-Led Intervention on Oral Health Among Hong Kong Adolescents: A Cluster-Randomized Controlled Trial. J Adolesc Health. 2022 Feb;70(2):267-274. doi: 10.1016/j.jadohealth.2021.08.001. Epub 2021 Sep 11. PMID 34521576

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT03694496/Prot_002.pdf
  • Informed Consent Form (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03694496/ICF_001.pdf